CLINICAL TRIAL: NCT05740033
Title: Functional and Aesthetic Outcomes of Radial Forearm Free Flap Closure Using Split-Thickness Skin Graft vs Primary Closure; a Randomized Control Trial
Brief Title: Radial Forearm Donor Site Closure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Eitan Prisman, Clinical Associate Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H22-02104
Record Dates: First submitted 2023-01-03; First posted 2023-02-22 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Oral Cancer; Oral Cavity Cancer; Donor Site Complication
Keywords: Oral Cancer; Oral Cavity Cancer; Radial Forearm; Donor Site; Surgical Complications
MeSH Terms: conditions — Mouth Neoplasms

STUDY DESIGN:
Intervention Model Description: The study will have two arms: one with participants receiving a split-thickness skin graft from the thigh to close the radial forearm donor site, and the other using a local (hatchet) flap to close this site. These two arms will be populated randomly and in parallel.
Masking Description: Participants will become aware of what arm they were randomly assigned to: those in the STSG arm will be to see their additional thigh scar; those in the local flap arm will lack this scar. As such, participants will only be blinded prior to their treatment. The surgeons may not be blinded as they will be performing the procedure on the participants and following up with them as per standard of care post-operatively.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- STSG arm (Active Comparator): Patient demographics will be recorded during the enrollment visit. During the participant's surgery in which the radial forearm free flap (RFFF) has been used, surgeons will perform a split-thickness thigh graft to close the forearm donor site. A photograph will be taken of the participants' forearm upon the removal of the dressing and splint.
  On each of the two follow-up clinic visits, another photo will be taken of the forearm scar and patient-reported outcome questionnaires will be provided for completion.
  Interventions: Procedure: Split-Thickness Skin Graft for Radial Forearm Donor Site Closure
- Hatchet flap arm (Active Comparator): Patient demographics will be recorded during the enrollment visit. The hatchet flap closure of the forearm donor site will be performed following the RFFF's usage. A photograph will be taken of the participants' forearm upon the removal of the dressing and splint.
  On each of the two follow-up clinic visits, another photo will be taken of the forearm scar and patient-reported outcome questionnaires will be provided for completion.
  Interventions: Procedure: Hatchet Flap for Radial Forearm Donor Site Closure

INTERVENTIONS:
Procedure: Split-Thickness Skin Graft for Radial Forearm Donor Site Closure — This method is performed by harvesting a 0.014-inch skin graft harvested from the anterolateral thigh on the side of the RFFF to reconstruct the forearm donor site. This skin graft is then used to cover the donor defect. The skin graft is sutured in place with 4-0 chromic suture, and a standard bolster dressing will be applied, and a partial splint will be left in place for five days post-operation.
  Arms: STSG arm
Procedure: Hatchet Flap for Radial Forearm Donor Site Closure — The hatchet flap closures will be performed based on prior description by Lane et al. (12), except no drain is placed in situ. A back cut of 3 to 4 cm is made to aid closure (Figure 1). Tension will be minimized by maintaining the wrist in flexion. A mepore dressing will be applied to the donor site post-operatively for two days.
  Arms: Hatchet flap arm

SUMMARY:
The radial forearm free flap (RFFF) is widely used in head and neck reconstruction. Its thinness, pliability, pedicle length, and vessel size are particularly suited for oropharyngeal and oral cavity reconstruction. Concerns about aesthetic and functional morbidity at the donor site have given rise to various techniques of closing the donor site, two of which are the split-thickness skin graft (STSG), taken from the thigh, and the hatchet flap, which uses a local flap within the radial forearm. This RCT will determine whether retrospectively reported improvements to aesthetic and functional outcomes for STSG patients are greater compared to hatchet flap patients.

DETAILED DESCRIPTION:
The radial forearm free flap (RFFF), introduced by Yang et al. in 1981, is widely used in head and neck reconstruction. Its thinness, pliability, pedicle length, and vessel size are particularly suited for oropharyngeal and oral cavity reconstruction. Since the survival rate of the RFFF has reached more than 95%, the clinical focus has gradually shifted to the postoperative quality of life, particularly in terms of donor site morbidity.

Concerns about aesthetic and functional morbidity at the donor site have given rise to various techniques of closing the donor site of a RFFF. Many possibilities of donor site closures have been described, ranging from direct closure to skin grafting, tissue expansion, use of acellular dermal matrix and local flaps. Each of these techniques has its own advantages and drawbacks and the debate regarding the optimal method for closing the RFFF donor site continues.

Split-thickness skin graft (STSG) is a very thin strip of skin that is typically taken from the upper thigh and is the most commonly used method to cover the forearm after taking the RFFF. Advantages of this technique include reducing the amount of tension that is on the forearm which may lead to a better scar and better mobility while disadvantages include the need of an additional scar on the thigh and possible mismatch of the color of the skin graft when compared to the forearm.

Due to these potential limitations, surgeons have attempted to close the forearm directly by means of local flaps, which use nearby skin, soft tissue, and blood vessels to cover the forearm. The hatchet flap is a triangular local rotation flap, first described by Emmet in 1977, with a greater or lesser degree of advancement and with a back cut at the base of the flap through which it derives its vascular supply. This method may allow for quicker wound healing by primary intention and improved coverage of the tendons which should theoretically decrease donor site morbidity; however, since only tissue from the forearm is used this may lead to increased tension and therefore increased scar formation.

Risks and complications for both types of closure are the same which include bleeding, infection, hypertrophic scars, tendon exposure, divot formation, irregular skin graft surface, prolonged wound healing, and loss of skin graft. There are only a few studies on the functional and visual outcomes of forearm closure after RFFF removal using the hatchet flap or similar local flaps, warranting the need for further studies on these closure techniques.

It is hypothesized that donor site closure using the STSG flap will result in greater functional and aesthetic outcomes for the radial forearm donor site as measured by an improved scores to the 3 given questionnaires. Post-operative complication rates are also hypothesized to be lower for STSG flap closure when compared to hatchet flap closure.

The literature currently remains in a state of clinical equipoise, and at the study site (Vancouver General Hospital) the STSG and hatchet flap are the two most common methods of donor site closure. Based on a retrospective data analysis at the study site, functional and patient-reported scar aesthetic outcomes were improved for STSG flap closure patients when compared to hatchet flap patients. As a retrospective analysis, objective assessments of the scar could not be performed, nor could the immediate post-operative outcomes be taken and compared over a consistent post-operative time frame schedule. This study aims to address this knowledge gap by conducting a parallel-group randomized controlled trial for the study site's two common donor site closure techniques, STSG and hatchet flap.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 or older
* Oral cavity disease (malignant or benign) requiring radial forearm free flap reconstruction

Exclusion Criteria:

* Serious medical comorbidities including metastatic disease or other contraindications to surgery
* Any pre-existing condition affecting the use of both hands, including previous major scars
* Unable or unwilling to complete post-operative questionnaires in English
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
First Michigan Hand Outcomes Questionnaire (MHOQ) Measure | Measure documented at 1 month post-surgery.
  A questionnaire that measures symptoms, function, aesthetics, and patient satisfaction in regards to the function of their hands. Responses are recorded on a 5-point Likert scale ranging from very good (1) to very poor (5).
Second MHOQ Measure | Measure documented between 3-6 months post-surgery.
  A questionnaire that measures symptoms, function, aesthetics, and patient satisfaction in regards to the function of their hands. Responses are recorded on a 5-point Likert scale ranging from very good (1) to very poor (5).
First Patient and Observer Scale Assessment Scale (POSAS) Measure | Measure documented at 1 month post-surgery.
  A questionnaire measuring both the patient's aesthetic perception and the trial coordinator's aesthetic and physical assessment of the scar formation along the donor site wound. Responses to questions are measured on a 10-point Likert scale ranging from the worst scarring imaginable (10) to the best scar imaginable (feels like normal skin, not scar tissue; 1).
Second POSAS Measure | Measure documented between 3-6 months post-surgery.
  A questionnaire measuring both the patient's aesthetic perception and the trial coordinator's aesthetic and physical assessment of the scar formation along the donor site wound. Responses to questions are measured on a 10-point Likert scale ranging from the worst scarring imaginable (10) to the best scar imaginable (feels like normal skin, not scar tissue; 1).
First Decision Regret Scale (DRS) Measure | Measure documented at 1 month post-surgery.
  A questionnaire measuring a patient's decisional regret related to receiving the surgery. Responses are measured on a 5-point Likert scale, ranging from extreme decisional regret (5) to no decisional regret (1).
Second DRS Measure | Measure documented between 3-6 months post-surgery.
  A questionnaire measuring a patient's decisional regret related to receiving the surgery. Responses are measured on a 5-point Likert scale, ranging from extreme decisional regret (5) to no decisional regret (1).

SECONDARY OUTCOMES:
Localized Hematoma at Donor Site | Patients will be monitored for 6 months post-operatively.
  A severe pooling of blood at the donor site.
Donor Site Infection | Patients will be monitored for 6 months post-operatively.
  Infection at the donor site or anywhere along the forearm scar.
Donor Site Wound Dehiscence | Patients will be monitored for 6 months post-operatively.
  A re-opening of the donor site wound.
Donor Site Tendon Exposure | Patients will be monitored for 6 months post-operatively.
  Exposure of the forearm tendons at the donor site.
Donor Site Skin Necrosis | Patients will be monitored for 6 months post-operatively.
  Significant amount of dead or dying skin tissue overlying or abutting the donor site and scar.
Donor Site Contractures | Patients will be monitored for 6 months post-operatively.
  A persistent tightening or contraction of skin, ligaments, tendons, or muscles at the forearm donor site.
Keloid Scarring at Donor Site Wound | Patients will be monitored for 6 months post-operatively.
  Excessive scar tissue formation along the donor site wound.
Divot Formation into Skin at Donor Site | Patients will be monitored for 6 months post-operatively.
  Visible and persistent depressions into the skin surface of the forearm.
Skin Graft Irregularities at Donor Site | Patients will be monitored for 6 months post-operatively.
  Additional irregularities such as bumps, roughness, or changes to colour will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada